CLINICAL TRIAL: NCT01139788
Title: A Phase 1 Study of LY2624587 in Patients With Advanced Cancer
Brief Title: A Study of LY2624587 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13740; I4N-MC-CXBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-27; First posted 2010-06-09 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Metastatic Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — LY2624587

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2624587 (Experimental)
  Interventions: Drug: LY2624587

INTERVENTIONS:
Drug: LY2624587 — 6-900 mg, administered intravenously, weekly for a minimum of one (1) 28 day cycle.
  If patients are determined to be receiving benefit, study treatment may be continued for up to one (1) year (12 cycles of 28 days).

SUMMARY:
Study CXBA is a multicenter nonrandomized, dose escalation, open-label, Phase 1 study of intravenous LY2624587 in patients with advanced or metastatic cancer for which no treatment of higher priority exists.

ELIGIBILITY:
Inclusion Criteria:

* Present with histological or cytological evidence of a diagnosis of cancer (solid tumors, lymphoma, or chronic lymphocytic leukemia) that is advanced and/or metastatic. The patient must be, in the judgement of the investigator, an appropriate candidate for experimental therapy after available standard therapies have been used.
* Have the presence of measurable or nonmeasurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST), Revised International Working Group Lymphoma Response Criteria, or National Cancer Institute Working Group Guidelines for Chronic Lymphocytic Leukemia.
* Have adequate organ function.
* Have a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug.
* Females with child bearing potential must have had a negative serum pregnancy test less than or equal to 7 days prior to the first dose of study drug.
* Have discontinued chemotherapy and cancer-related hormonal therapy with commercially-available agents for at least 21 days (6 weeks for mitomycin-C or nitrosoureas) and radiotherapy for at least 14 days prior to study enrollment and recovered from the acute effects of therapy (less than or equal to National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE v 4.02; Grade 1). Hormone refractory prostate cancer patients receiving gonadotropin releasing hormone (GnRH) agonist therapy or breast cancer patients on anti-estrogen therapy (for example, an aromatase inhibitor) prior to entrance on the study may have that treatment continued while they are enrolled in Study CXBA.
* Have an estimated life expectancy of greater than or equal to 12 weeks.

Exclusion Criteria:

* Have received treatment with an investigational drug, which has not received regulatory approval for any indication, within 28 days of study treatment with LY2624587.
* Have medical conditions that, in the opinion of the investigator, would preclude participation in this study.
* Have symptomatic central nervous system malignancy or metastasis. Patients with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic patients without history of CNS metastases is not required.
* Have a history of major organ transplant.
* Have current acute leukemia.
* Have active human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C antibodies.
* Have QTc greater than 470 msec (female) or greater than450 msec (male), history of congenital long QT syndrome or other conduction abnormality.
* Have had an autologous or allogenic bone marrow transplant.
* Previously treated with a CXCR4 antagonist, or have had a significant allergy to biologic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Recommended dose for Phase 2 studies | Baseline to study completion

SECONDARY OUTCOMES:
Number of participants with clinically significant effects | Baseline to cycle 12
Radiological tumor measurement | Baseline, Cycle 1 Day-1, Cycle 2 - Day 1, Cycle 3 - Day 1
Pharmacokinetics of LY2624587, area under the concentration-time curve (AUC) | Cycle 1 - Cycle 12
Pharmacodynamic, maximum peak concentration (Cmax). | Baseline to date last subject discontinues from study drug

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hour EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas